CLINICAL TRIAL: NCT05892887
Title: Analgesic Efficacy of Different Volumes in Erector Spinae Plane Block in Patients Undergoing Single Level Lumbar Spine Fixation: A Non-inferiority Randomized Clinical Trial
Brief Title: Analgesic Efficacy of Different Volumes in Erector Spinae Plane Block in Single Level Lumbar Spine Fixation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Kafrelsheikh University, Kafrelsheikh, Egypt, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 50- 1 - 10
Record Dates: First submitted 2023-05-10; First posted 2023-06-07 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Erector 10 (Experimental): Received 10ml of preoperative bilateral ultrasound guided ESPB by bupivacaine 0.25% on each side
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Erector 15 (Experimental): Received 15ml of preoperative bilateral ultrasound guided ESPB by bupivacaine 0.25% on each side
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Erector 20 (Experimental): Received 20ml of preoperative bilateral ultrasound guided ESPB by bupivacaine 0.25% on each side
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — Bilateral ultrasound guided in erector spinae plane block by bupivacaine 0.25%

SUMMARY:
The analgesic efficacy of different volumes in ESPB patients undergoing single-level lumbar spine fixation

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) its an interfacial plane block for an effective treatment for thoracic neuropathic pain. Currently, compared to the use of opioids, the ESPB has fewer side effects and is safe for patients of all ages having abdominal and thoracic operations .

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years.
2. Both genders.
3. American Society of Anesthesiologists' (ASA) physical status I or II.
4. Undergoing single level lumbar spine fixation.

Exclusion Criteria:

1. Patient refusal.
2. Pregnant females.
3. Renal, lung, heart, or liver disorders.
4. Communication difficulties which might prevent a reliable postoperative assessment.
5. Contraindication to regional anesthesia (bleeding disorder, use of any anticoagulants, local infection, known allergy to local anesthetics).
6. BMI more than 30 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | First 24 hours postoperatively
  Patients were allowed to receive incremental doses of morphine 3mg intravenously if numerical rating scale pain score will be ≥ then the total amount of morphine will be recorded

SECONDARY OUTCOMES:
Numerical rating scale | Up to 48 hours postoperatively
  Postoperative pain using numerical rating scale (NRS) will be measured at post-anesthesia care unit, from 0 to 10, with 0 representing no pain and 10 representing maximum intolerable pain
Time to the first rescue analgesic | Up to 24 hours postoperatively
  If numerical rating scale >4 was observed, rescue analgesia (morphine 3 mg IV) was administered
Postoperative complications | Up to 24 hours postoperatively
  postoperative nausea and vomiting (PONV), hypotension (mean arterial pressure < 20% of baseline readings and was managed by ephedrine 5 mg IV and/or normal saline IVI), bradycardia (heart rate < 60 beats/min and was managed by atropine 0.6 mg IV).
5-point scale | Up to 24 hours postoperative
  The degree of patient satisfaction was assessed on a 5-point scale: (0= extremely dissatisfied, 1= unsatisfied, 2= neither satisfied nor unsatisfied, 3= satisfied), and 4= extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: The data will be available after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Algyar MF, Zahra AA, Elshikhali AS, Abdelhameed EA, El Hefny DA, Moharam SA, ElSharkawy MS, Farghaly OS, Ahmed MA. Analgesic efficacy of different volumes in erector spinae plane block in patients undergoing single level lumbar spine fixation: a non-inferiority randomized trial. BMC Anesthesiol. 2025 Sep 1;25(1):439. doi: 10.1186/s12871-025-03247-z. PMID 40890575